CLINICAL TRIAL: NCT02435030
Title: A Prospective Non-therapeutic Study in Patients Diagnosed With Niemann-Pick Disease Type C in Order to Characterise the Individual Patient Disease Profile and Historic Signo-symptomatology Progression Pattern
Brief Title: A Prospective Non-therapeutic Study in Patients Diagnosed With Niemann-Pick Disease Type C
Status: Completed | Type: Observational
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-ORZY-NPC-001; 2014-005194-37 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: NP-C; LSD; lysosomal storage disorder; lysosomal storage disease; NPC2; NPC1; Niemann-Pick Type C; Niemann-Pick,; Arimoclomol
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NP-C Patients: NPC type 1 or 2 patients aged 2-18 years

SUMMARY:
This is a prospective non-therapeutic observational study in NP-C patients. The aim is to characterize the individual patient disease progression profile through the historical and 6 months prospective evaluation of clinical, imaging, biological(biomarkers) and quality of life data.

Patients will be offered enrollment into a Phase II/III study on arimoclomol at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent if appropriate to local laws and regulations) prior to any study-related procedures;
* Males and females aged from 2 years to 18 years and 11 months;
* Patients of any ethnic background will be eligible for this study;
* Patient weight ≥15th percentile of body mass index (BMI) for age according to the World Health Organisation (WHO) standards;
* Diagnosis of Niemann Pick disease Type C (NP-C), either NPC1 or NPC2;
* NP-C diagnosis genetically confirmed (deoxyribonucleic acid [DNA] sequence analysis);
* Both NPC1 and NPC2 patients are eligible;
* Presenting at least one neurological symptom of the disease (for example, but not limited to, hearing loss, vertical supranuclear gaze palsy, ataxia, dementia, dystonia, seizures, dysarthria, or dysphagia);
* Ability to walk either independently or with assistance;
* Ability to travel to the corresponding clinical trial site repeatedly (every 6 months) for evaluation and follow-up;
* Treated or non-treated with miglustat;
* If a patient is under prescribed treatment with miglustat, it has to be under stable dose of the medication for ≥ 3 continuous months prior to inclusion in the study;
* Sexually active patients must be willing and able to use an adequate method of contraception throughout the study, for example: diaphragm + spermicide; intrauterine contraceptive device; oral contraceptives; implant; injection of a progestogen medication;
* Ability to comply with the protocol-specified procedures/evaluations and scheduled visits;
* Willing to participate in all aspects of trial design including serial blood sampling, skin biopsies and imaging (ultrasonography) collections.

Exclusion Criteria:

* No written informed consent obtained from the patient or their parent(s)/legal guardian(s) (and assent if appropriate to local laws and regulation) before any study related procedures;
* Recipient of a liver transplant or planned liver transplantation;
* Patients with uncontrolled severe epileptic seizures period (at least 3 consecutive severe epileptic seizures that required medication) within 2 months prior to the written consent. This includes patients with ongoing seizures that are not stable in frequency or type or duration over a 2 month period prior to enrollment, requiring change in dose of antiepileptic medication (other than adjustment for weight) over a 2 month period prior to enrollment, or requiring 3 or more antiepileptic medications to control seizures;
* Neurologically asymptomatic patients;
* Severe liver insufficiency (defined as hepatic laboratory parameters, aspartate transaminase [AST] and alanine transaminase [ALT] greater than three-times the upper limit of normal for age and gender;
* Severe renal insufficiency, with serum creatinine level greater than 1.5 times the upper limit of normal ;
* Severe manifestations of NP-C disease that would interfere with the patient's ability to comply with the requirements of this protocol;
* In the opinion of the Investigator, the patient's clinical condition does not allow for the required blood collection and/or skin biopsies as per the protocol-specified procedures;
* Treatment with any IMP within 4 weeks prior to the study enrollment;
* Treatment with any IMP during the study in an attempt to treat NP-C;
* Current participation in another trial is not permitted unless it is a non-interventional study and the sole purpose of the trial is for long-term follow up/survival data (registry);
* Patients will be excluded if there is a confirmed risk linked to the MRI procedure to be performed in the subsequent therapeutic interventional study [i.e.: implanted cardiac pacemaker or implantable cardioverter defibrillator, implanted neural pacemakers, cochlear implants, implanted metallic foreign bodies in the eye or CNS (such as a CNS aneurysmal clip), any form of implanted wire or metal device that may concentrate radio frequency fields and/or confirmed history of unexpected serious adverse reaction to sedation or anesthesia (if sedation is necessary)];
* Patients will be excluded if there is a confirmed risk linked to the skin punch biopsy procedure like severe thrombocytopaenia, at investigator's discretion.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: NPC1 and NPC2 patients aged 2-18 years
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
NP-C clinical disease severity | at week 0 and week 24-28
  Change in NP-C Clinical Severity scale
Quality of life questionnaire (EQ-5D-Y) | at week 0 and week 24-28
  Change in the Quality of life
Ultrasonographic evaluation of liver and spleen | at week 0 and week 24-28
  Changes in the size and/or characteristics of the liver and spleen (assessed by ultrasound).
Oxysterol | at week 0 and week 24-28
  Change in Oxysterol concentrations
NPC clinical symptoms | at week 0 and week 24-28
  Change in NPC clinical symptoms
NPC protein | at week 0 and week 24-28
  Change in NPC protein concentrations

SECONDARY OUTCOMES:
Safety Parameters | at week 0 and week 24-28
  Adverse events (AEs) (disease related and treatment related), haematology, clinical chemistry, physical examination, vital signs and electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Eugen Mengel, Principal Investigator — Villa Metabolica, Mainz, Germany
Locations (16):
- University Hospital Copenhagen (Rigshospitalet), Copenhagen, Denmark
- France (2):
  - CHU de Montpellier, Montpellier
  - Hôpital Trousseau, Paris
- Germany (2):
  - Villa Metabolica Mainz, Mainz
  - Klinikum der Universistat, Munchen, Munich
- Italy (5):
  - Istituto Carlo Besta (Milano), Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Università Federico II, Napoli
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine
- The Children´s Memorial Istitute Warsaw, Warsaw, Poland
- Spain (2):
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Quirón, Zaragoza
- Inselspital, University Hospital Bern, Bern, Switzerland
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital, London

REFERENCES:
- [Derived] Mengel E, Bembi B, Del Toro M, Deodato F, Gautschi M, Grunewald S, Gronborg S, Heron B, Maier EM, Roubertie A, Santra S, Tylki-Szymanska A, Day S, Symonds T, Hudgens S, Patterson MC, Guldberg C, Ingemann L, Petersen NHT, Kirkegaard T, I Dali C. Clinical disease progression and biomarkers in Niemann-Pick disease type C: a prospective cohort study. Orphanet J Rare Dis. 2020 Nov 23;15(1):328. doi: 10.1186/s13023-020-01616-0. PMID 33228797